CLINICAL TRIAL: NCT07378202
Title: Machine Learning for Prediction of Therapy Response in Autoimmune Hepatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Engel, Bastian Dr., Gastroenterologist, Clinician Scientist, Principal Investigator, Hannover Medical School
Other Study IDs: AIH_ML_v1
Record Dates: First submitted 2026-01-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Hepatitis
Keywords: machine learning; registry; therapeutic response
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- R-LIVER Registry
- AIH registry from Edmonton, Canada
- CANAL Registry
- IAIHG Registry
- ColHAI Registry

SUMMARY:
The 5th International Autoimmune Hepatitis Group (IAIHG) research workshop emphasized the integration of large clinical cohorts with artificial intelligence (AI) for enhanced prediction of therapy responses and outcomes in Autoimmune Hepatitis (AIH). This project aims to develop and validate machine learning (ML) models using data from the R-Liver registry and other international cohorts. After rigorous preprocessing to ensure data uniformity and quality, the investigators will identify and characterize factors influencing therapy response. They will then implement ML models to predict complete biochemical response (CBR) at 6 and 12 months, using five-fold cross-validation, and validate these models in external cohorts from Spain, Canada, and the international AIH group, ensuring robustness and generalizability.

Finally, the investigators will prospectively validate the models in newly registered cases, assessing both short-term and long-term outcomes. This project seeks to advance personalized treatment strategies in AIH, facilitating timely adjustments in therapy and improving patient prognosis through AI-driven decision support. This projects' interdisciplinary team, with expertise in clinical AI and hepatology, is well-equipped to address these challenges and enhance the clinical management of AIH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autoimmune hepatitis
* Consent to provide data to the specific registry
* available follow-up data at least within the first 12 months

Exclusion Criteria:

* variant syndromes
* extrahepatic autoimmune disease
* immunosuppressive treatment at diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This project utilizes already established registries of patients with autoimmune hepatitis (AIH) from the international autoimmune hepatitis group (IAIHG), the European Reference Network on Rare liver diseases (R-LIVER), the spanish network on autoimmune hepatitis (colHAI) and the canadian network on autoimmune hepatitis (CANAL). Initial reports on the patient populations within the respective registries were separately published (doi: 10.1111/liv.16035, doi: 10.1097/HEP.0000000000000589, 10.1016/j.jhep.2024.03.021, 10.1097/HEP.0000000000000018 ).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete biochemical response at 6 months after diagnosis | 6 months
  Complete biochemical response is defined as normal aspartate amino transferase (AST), alanine aminotransferase (ALT) and immunoglobulin G (IgG).
Number of patients with complete biochemical response at 12 months after diagnosis | 12 months
  Complete biochemical response is defined as normal aspartate amino transferase (AST), alanine aminotransferase (ALT) and immunoglobulin G (IgG).

SECONDARY OUTCOMES:
Number of patients experiencing liver-related death or liver transplantation | From enrolment until the end of the study
Number of patients with decompensation of liver disease | From enrolment until the end of the study
  Decompensation meaning a composite of new/worsening ascites, infection requiring hospitalization, acute-on-chronic liver failure, variceal bleeding, hepatic encephalopathy.
Number of patients with complete biochemical response through study completion | through study completion, an expected average of 1 year
  Complete biochemical response is defined by normal AST, normal ALT and normal IgG
Number of patients with histological remission of AIH through study completion | through study completion, an expected average of 1 year
  Histological remission is defined as modified hepatitis activity index below 4.
Number of patients that develop cirrhosis through study completion | through study completion, an expected average of 1 year
  Cirrhosis is defined by imaging findings indicative of cirrhosis, histological staging indicating fibrosis or liver stiffness measurement that is in line with a cirrhotic liver.
Number of patients with intolerance to primary treatment necessitating regimen change | 12 months
  Intolerance to treatment is reported by respective patients and assessed by respective treating physicians. It is expected to be gastrointestinal side effects and hematological side effects (cytopenias) that may typically occur from treatment with azathioprine or mycophenolate mofetil which lead to change of treatment regimens in patients with autoimmune hepatitis.
Number of patients with non-response to primary treatment necessitating treatment change | 12 months
  Non-Response ist defined as persistently elevated aspartate aminotransferase, alanine aminotransferase and/or immunoglobulin G. It is considered a reason to change the therapeutic regimen.
Number of patients with third line treatment due to non-response to obtain biochemical response through study completion | through study completion, an expected average of 1 year
  Non-response is defined as persistently elevated aminotransferases and/or immunoglobulin G.
Number of patients with normalization of aminotransferase levels in the blood irrespective of Immunoglobulin G levels | 6 months
  Aminotransferases are alanine aminotransferase and asparatate aminotransferase. These enzymes indicate liver injury and are considered response markers measured from blood in clinical routine to assess therapeutic response in autoimmune hepatitis.
Number of patients with normalization of aminotransferase levels irrespective of Immunoglobulin G levels | 12 months
  Aminotransferases are alanine aminotransferase and asparatate aminotransferase. These enzymes indicate liver injury and are considered response markers measured from blood in clinical routine to assess therapeutic response in autoimmune hepatitis.
Number of patients with steroid-free complete biochemical response | 6 months
  Complete biochemical response is defined by normal blood levels for aminotransferases and normal immunoglobulin G. This outcome measure assesses this parameter in relation to the fact if the patient needed corticosteroid-therapy to obtain this outcome or if the patient only needed other immunosuppressive drugs (e.g. azathioprine, mycophenolate mofetil).
Number of patients with steroid-free complete biochemical response | 12 months
  Complete biochemical response is defined by normal blood levels for aminotransferases and normal immunoglobulin G. This outcome measure assesses this parameter in relation to the fact if the patient needed corticosteroid-therapy to obtain this outcome or if the patient only needed other immunosuppressive drugs (e.g. azathioprine, mycophenolate mofetil).

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Engel, MD, Principal Investigator — Hannover Medical School, Hannover, Germany
Locations (2):
- Germany (2):
  - Else Kroener Fresenius Center for Digital Health, Technical University Dresden, Dresden
  - Hannover Medical School, Hanover

IPD SHARING:
Plan to Share IPD: No
Anonymized IPD will be shared for the purpose of the study by the respective registries with the research team of this study. IPD request need to be directed directly to the respective officials of the different registries.